CLINICAL TRIAL: NCT02098304
Title: Post-Approval Clinical Study to Evaluate the Safety and Performance of the Calcivis Caries Activity Imaging System in a Clinical Setting
Brief Title: Post-Approval Clinical Study to Evaluate the Calcivis Caries Activity Imaging System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calcivis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CAL-01-2013
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-03

CONDITIONS: Dental Caries
Keywords: Caries; ICDAS; Lesion activity; Demineralisation; Imaging
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sound and Unsound Molars (Other): Imaging of unrestored sound molars (ICDAS 0), and third Molars (ICDAS 1,2 or 3) with the Calcivis Caries Activity Imaging System
  Interventions: Device: Calcivis Caries Activity Imaging System

INTERVENTIONS:
Device: Calcivis Caries Activity Imaging System — Teeth imaged with the Calcivis Caries Activity Imaging System

SUMMARY:
This is a prospective, multi-centre, post-approval clinical study to assess the safety and the performance of the Calcivis Caries Activity Imaging System in aiding the identification of active caries lesions on the occlusal surfaces of human teeth. Following the identification of potential caries lesions by oral examination under ICDAS (International Caries Detection and Assessment System) guidelines, a disclosing solution will be applied which will cause areas of active demineralization (loss of calcium ions) to luminesce - these will be captured with an intra-oral camera to produce mapping images of the tooth surface. For the purposes of this study the presence / absence of luminescence will be used as an indicator of lesion activity / inactivity.

The study will be deemed a success if the level of agreement between elevated luminescence with the Calcivis System, and areas of expected lesion activity as rated by the Investigators ICDAS staging, is above 70%, is not due to chance and correlates well with published data on active non-cavitated lesions in molars at various stages of eruption.

DETAILED DESCRIPTION:
Dental caries (tooth decay) is a significant clinical and public health problem. The development of caries lesions involves a net mineral loss of dental tissue, which can lead to progressive loss of tooth structure surface, associated pain and disease. Detecting, assessing, diagnosing and treating such lesions are core activities in dentistry. Currently the main detection and diagnosis aids are visual inspection and the use of a probe, together with X-ray images. Determination of the activity status of a lesion (how likely it is to progress) is required to assess treatment needs. Currently methods are problematic and involve the clinician's subjective assessment and / or monitoring lesion progression over a number of visits.

Therefore, this prospective, multi-centre, post-approval clinical study has been designed to assess the safety and performance of the Calcivis Caries Activity Imaging System in a clinical setting.

The device under evaluation - the Calcivis Caries Activity Imaging System comprises a hand-held specialised intra-oral camera which takes images of the lesion on the tooth surface immediately before and after application of a disclosing solution which contains a photoprotein. This photoprotein will detect free calcium ions on the tooth surface and produces a visible light signal if the caries lesion is active.

Patients attending routine dental appointments and / or patients on the dental practice register, who are identified by the Investigator as meeting all the study inclusion and exclusion criteria will be approached to discuss their possible participation in the study. Patients will be given a Patient Information Sheet to read and time to consider their participation. If they agree to participate, they will be asked to attend for two study visits, one week apart. Written informed consent will be taken before any study procedures are conducted.

At Study Visit 1, pre-imaging demographics and oral hygiene information will be collected. All occlusal surfaces of the teeth (12 possible molars and pre-molars) will be cleaned by the Dentist, by brushing with dental paste and rinsing with tap water and using a 3-in-1 air / water spray, according to a Tooth Cleaning Protocol. The Dentist will then perform an oral examination identifying and noting the ICDAS score of each tooth to be imaged with the Calcivis System. Colour photographs will be taken with a standard intra-oral camera of each selected molar and surrounding mucosa. Each tooth selected for imaging will be air dried for 5 seconds immediately before application of the disclosing solution and imaging. Images of one sound tooth and one unrestored erupted, or erupting third molar with an ICDAS score of 1,2 or 3 will be imaged. An additional two teeth may be imaged (remaining erupted / erupting third molar and / or any other molar with an ICDAS score of 1,2 or 3), up to a maximum of four teeth. Immediately after imaging has been completed, patients rinse out with tap water and a second colour photograph will be taken with a standard intra-oral camera of each selected molar and surrounding mucosa. Any adverse events will be recorded.

Post-imaging Questionnaires will be completed by all patients at the end of Study Visit 1, and User Questionnaires will be completed at the end of each Study Visit day.

Patients will return after one week for Study Visit 2. At this visit, a final oral examination will be conducted and colour will be taken with a standard intra-oral camera of each selected molar and surrounding mucosa. Any adverse events observed or volunteered by the patient will be recorded.

At the end of either Study Visit 1 or 2, the Dentist may share the images of the teeth imaged with the Calcivis System with the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 16 to 25 years old
2. Patient must have at least one unrestored molar identified as sound according to the ICDAS coding system
3. Patient must have at least one unrestored erupting (in which case occlusal surface must be such that, apart from minimal presence of an operculum over the distal marginal ridge, it is clear of the gingivae (gum)) or erupted third molar with a caries lesion identified, coded 1, 2 or 3 (according to the ICDAS coding system)
4. Patient must be willing and able to give written informed consent
5. Patient must be willing and able to adhere to study schedule

Exclusion Criteria:

1. Recent tooth bleaching (within previous two weeks of imaging with the Calcivis System)
2. On-going re-mineralisation treatment including, but not limited to high concentration prescription fluoride toothpaste
3. Any patient with a fixed orthodontic appliance
4. Any patient currently taking part in a clinical research study, or has taken part in a clinical research study in the previous three months
5. Pregnant and / or nursing mothers

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ormond, BDS,MGDS,FDS, Principal Investigator — Clark and Watson Dental Practice
Locations (3):
- United Kingdom (3):
  - Bathgate Smile Centre, Bathgate
  - Downie, Haper and Shanks Dental Practice, Edinburgh
  - Clark and Watson Dental Practice, Falkirk

IPD SHARING:
Plan to Share IPD: Yes
Final Clinical Study Report issued

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 Patients were recruited to the study from three UK General Dental Practices by four investigators. All 42 patients attended both Visit 1 and 2 and completed the study. There were no patient withdrawals. Patients were recruited at the three sites over an 8 month period from May 2014 to January 2015.
Groups:
- Sound and Unsound Molars: Imaging of unrestored sound molars (ICDAS 0) and third molars (ICDAS 1,2 or 3) with the Calcivis Caries Activity Imaging System
Period: Overall Study
Arm/Group | Sound and Unsound Molars
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients were recruited who had at least one unrestored molar identified as sound AND at least one unrestored erupting or erupted third molar coded ICDAS 1,2 or 3.
Groups:
- Sound and Unsound Molars: Imaging of unrestored sound molars (ICDAS 0) and third Molars (ICDAS 1,2 or 3) with the Calcivis Caries Activity Imaging Device
  Calcivis Caries Activity Imaging System: Unrestored sound molars and unsound molars imaged with the Calcivis Caries Activity Imaging System
Arm/Group | Sound and Unsound Molars
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 21.7 [17 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 42
  Black African | 0
  Asian | 0
  Hispanic | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage Agreement of Sound/Unsound Teeth Between ICDAS Score and Calcivis System
Description: % agreement calculated as no. of teeth where ICDAS assessment & Calcivis System assessment is in agreement/total number of teeth assessed multiplied by 100. Agreement defined as a sound tooth without luminescence & an unsound tooth with luminescence.
Time Frame: Day 0
Population: All 42 patients recruited are included in the Safety Population, which included any subjects on whom the Calcivis System was used. 31 patients are included in the Agreement Population which included all subjects with at least one tooth with an eligible image. From the 31 patients, 65 teeth were analysed; in some patients multiple teeth were imaged.
Measure: Number (95% Confidence Interval); unit: percentage agreement
Units Other Than Participants: teeth
Groups:
- Sound and Unsound Molars: Imaging of unrestored sound molars (ICDAS 0) and third molars (ICDAS 1, 2 or 3) with the Calcivis Caries Activity Imaging System
Arm/Group | Sound and Unsound Molars
Number analyzed (Participants) | 31
Number analyzed (teeth) | 65
percentage agreement | 72.3 [59.8 to 82.7]
Statistical Analysis 1: Comparison: Sound and Unsound Molars; The null hypothesis was of chance agreement (50%) and was tested against a two-sided alternative at the 5% level of significance; Test type: Superiority or Other; p < 0.001, Exact binomial test; An exact binomial test was used and an exact 95% Confidence Interval using the Clopper-Pearson method was calculated; Percentage agreement = 72.3, 95% CI 2-sided [59.8 to 82.7]
Statistical Analysis 2: Comparison: Sound and Unsound Molars; The null hypothesis was of chance agreement (Cohen's kappa of 0) and was tested against a two-sided alternative at the 5% level of significance. The study was powered such that 58 teeth (29 subjects), there would be 95% power to reject the null hypothesis of chance agreement (Cohen's kappa of 0) at the 5% level of significance, given that it was expected to be at least 0.4; Test type: Superiority or Other; p = 0.001, Cohen's Kappa; Cohen's kappa = 0.45, 95% CI 2-sided [0.24 to 0.66] — Cohen's kappa is a chance-adjusted measure of agreement. A value of 0 indicates agreement by chance and 1 perfect agreement

2. Primary Outcome: Measure Safety of the Calcivis Caries Imaging System
Description: Collection of all adverse events recorded and reported throughout the duration of the study
Time Frame: Day 0 and Day 7
Population: Adverse events
Measure: Number; unit: adverse events
Groups:
- Sound and Unsound Molars: Imaging of unrestored sound molars (ICDAS 0) and third Molars (ICDAS 1,2 or 3) with the Calcivis Caries Activity Imaging System
  Calcivis Caries Activity Imaging System: Unrestored sound molars and third molars imaged with the Calcivis Caries Activity Imaging System
Arm/Group | Sound and Unsound Molars
Number analyzed (Participants) | 42
adverse events | 2

3. Secondary Outcome: Patient Experience
Description: Completion of Patient Questionnaires after imaging with the Calcivis System
Time Frame: Day 0
Population: Patient Questionnaires comprised five questions and the patient was asked to tick the most appropriate response i.e very good, good etc. No numerical values were assigned to the responses
Measure: Number; unit: Patient Questionnaires
Units Other Than Participants: Patient Questionnaires
Arm/Group | Sound and Unsound Molars
Number analyzed (Participants) | 42
Number analyzed (Patient Questionnaires) | 42
Patient Questionnaires
  Overall experience with Calcivis System:very good | 30
  Overall experience with Calcivis System:good | 9
  Overall exp. with Calcivis System: not good or bad | 2
  Overall experience with Calcivis System: bad | 1
  Overall experience with Calcivis System: very bad | 0
  Overall exp. with Calcivis system: not recorded | 0
  Image review with Dentist: very helpful | 21
  Image review with Dentist:Helpful | 16
  Image review with Dentist:not helpful or unhelpful | 2
  Image review with dentist: unhelpful | 0
  Image review with Dentist: very unhelpful | 0
  Image review with Dentist: not recorded | 3
  Any pain from Calcivis System use: none | 34
  Any pain from Calcivis System use: slight | 5
  Any pain from Calcivis System Use: moderate | 2
  Any pain from Calcivis System use: marked | 1
  Any pain from Calcivis System use: severe | 0
  Any pain from Calcivis System use: not recorded | 0
  Any discomfort from Calvisi System use: none | 23
  Any discomfort from Calcivis System use: minor | 17
  Any discomfort from Calcivis System use: moderate | 1
  Any discomfort from Calcivis System use: marked | 1
  Any discomfort from Calcivis System use:severe | 0
  Any discomfort with Calcivis System: not recorded | 0
  Allow Calcivis System use in future: very happy | 35
  Allow Calcivis System use in furture: probably | 7
  Allow Calcivis System use in future: not sure | 0
  Allow Calcivis System use in future: possibly | 0
  Allow Calcivis System use in future: not allow | 0
  Allow Calcivis System use in future: not recorded | 0

4. Secondary Outcome: User Experience
Description: Completion of User Questionnaires after imaging with the Calcivis System
Time Frame: 0 day
Population: User Questionnaires comprised nine questions and users were asked to tick the most appropriate response i.e. extremely easy, easy etc. No numerical values were assigned to the responses.
Measure: Number; unit: User questionnaires
Arm/Group | Sound and Unsound Molars
Number analyzed (Participants) | 17
User questionnaires
  Calcivis System software use:extremely easy | 4
  Calcivis System software use:somewhat easy | 10
  Calcivis System software use:not easy or difficult | 2
  Calcivis System software use:somewhat difficult | 1
  Calcivis System software use:extremely difficult | 0
  Calcivis System software use:not recorded | 0
  Disclosing Solution preparation:extremely easy | 6
  Disclosing Solution preparation:somewhat easy | 7
  Disclosing Solution prep:not easy or difficult | 3
  Disclosing Solution prep:somewhat difficult | 1
  Disclsoing Solution prep.extremely difficult | 0
  Disclosing Solution prep:not recorded | 0
  Syringe loading & fit applicator:extremely easy | 6
  Syringe loading & fit applicator: somewhat easy | 9
  Syringe load & fit applicator:not easy ordifficult | 1
  Syringe load & fit applicator:somewhat difficult | 1
  Syringe load & fit applicator:extremely difficult | 0
  Syring load & fit applicator:not recorded | 0
  Device priming: extremely easy | 7
  Device priming: somewhat easy | 10
  Device priming: neither easy or difficult | 0
  Device priming: somewhat difficult | 0
  Device priming: extremely difficult | 0
  Device priming: not recorded | 0
  Ease of use of the device: extremely easy | 1
  Ease of use of the device:somwehat easy | 5
  Ease of use of the device: not easy or difficult | 1
  Ease of use of the device: somewhat difficult | 6
  Ease of use of the device: extremely difficult | 3
  Ease of use of the device: not recorded | 1
  Removal of applicator from device:extremeley easy | 12
  Removal of appliator from device: somewhat easy | 4
  Removal of applicator:not easy or difficult | 1
  Removal of applicator:somewhat difficult | 0
  Removal of applicator:extremely difficult | 0
  Removal of applicator: not recorded | 0
  Ease of cleaning device:extremely easy | 15
  Ease of cleaning device:somewhat easy | 1
  Ease of cleaning device:not easy or difficult | 0
  Ease of cleanig device:somewhat difficult | 0
  Ease of cleaning device:extremely difficult | 0
  Ease of cleaning device:not recorded | 1
  Overall experience with Calcivis System:very good | 0
  Overall experience with Calcivis System:good | 11
  Overall exp. with CS:not good or unsatisfactory | 2
  Overall exp. with CS:unsatisfactory | 2
  Overall exp.withCalcivis System:veryunsatisfactor | 1
  Overall exp. with Calcivis System:not recorded | 1
  Were IFU sufficient to understand:sufficient | 14
  Were IFU sufficient:somewhat sufficient | 1
  Were IFU sufficient:not sufficient or insufficient | 0
  Were IFU sufficient:somewhat insufficient | 0
  Were IFU sufficient to understand:insufficient | 0
  Were IFU sufficient to understand:not recorded | 2

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Sound and Unsound Molars
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sound and Unsound Molars (N=42)
Minor gum abrasion (Skin and subcutaneous tissue disorders) | 1 (1) — Minor gum abrasion to oral mucosa surrounding tooth
Bleeding gums (Skin and subcutaneous tissue disorders) | 1 (1) — Bleeding gums at margin of tooth and gums

LIMITATIONS AND CAVEATS:
All 42 patients recruited to the study are included in the Safety Population, however only 31 patients were included in the Agreement Population as one or more of the images from the Calcivis System were deemed ineligible by independent review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will not suppress or veto publications however the Sponsor reserves the right to postpone publication and/or communication for a short time to protect intellectual property.